CLINICAL TRIAL: NCT00497952
Title: Allogeneic Stem Cell Transplantation for the Treatment of Multiple Sclerosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: all clinical development programs terminated by sponsor
Sponsor: Talaris Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-13080-122206
Expanded Access: NCT02084121 (No longer available)
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing-remitting multiple sclerosis; Marrow/Stem cell transplant
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple Sclerosis Patients (Experimental): Recipients treated with a hematopoetic stem cell infusion from a living donor
  Interventions: Biological: hematopoetic stem cell infusion

INTERVENTIONS:
Biological: hematopoetic stem cell infusion — Enriched hematopoietic stem cell infusion

SUMMARY:
The goal of this research study is to establish chimerism with the goal to halt disease progression in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
While the cause of MS in not known, there is an autoimmune component that destroys nerve cells. Autoimmunity is a condition where an individual's immune system attacks his/her own cells. Bone marrow stem cell transplantation has been shown to halt autoimmunity. Stem cell transplant can be performed using the patient's own cells, or donor cells. The general consensus in the field is that donor transplant is most likely to halt disease progression. This study is designed to evaluate the safety of a donor transplant procedure as a therapy for relapsing remitting multiple sclerosis (RRMS).

Two factors limit the widespread application of traditional donor stem cell transplant: 1) preparing the patient for transplant (conditioning); and 2) graft-versus-host disease (GVHD). Traditional conditioning destroys the recipient's immune system and requires that the marrow transplant be successful because the patient is unable to fight off infection if the donor cells do not survive. GVHD occurs when donor immune cells recognize the recipient's cells as foreign tissue and attack them. Severe GVHD can result in death. This study utilizes a new approach to conditioning which leaves the patient's immune system intact. The transplant product is depleted of GVHD-producing cells but retains tolerance-promoting cells, called facilitating cells, which are intended to ensure the donor and recipient cells coexists peacefully. The toxicity of conditioning and transplantation is significantly reduced. The end result is a marrow system that contains recipient and donor cells, a state called mixed chimerism.

In this study, we will determine the appropriate cell dose to safely establish mixed chimerism following partial conditioning in patients with RRMS. The study takes a gradual approach to increasing the cell dose to achieve mixed chimerism. Each patient will receive a cell dose one unit above the dose received by the most recent safely transplanted patient. We believe this study will provide a breakthrough in the treatment of MS. The goal of this study is to evaluate the potential of safely establishing mixed chimerism to interrupt the autoimmune process and end the devastating effects of MS.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS according to the McDonald criteria
* Confirmed diagnosis of relapsing-remitting MS.
* Age between 18 and 55 years
* Extended Disability Status Score (EDSS) between 0 and 5.0
* Independently ambulatory (eligible for inclusion if subject was acutely non-ambulatory within the previous year and return of function is substantiated with EDSS score.)
* Relapse within the last year or sustained disability progression of 1.0 for six months
* Treatment with high dose, high frequency Interferon-β therapy, or failure to tolerate Interferon-β therapy
* Diffusing capacity of the lung for carbon monoxide (DLCO)> 50% (unless cleared by physician)
* Ejection fraction (EF) > 40% (unless cleared by cardiologist)
* Required initial laboratory data (obtained within 30 days prior to transplant, unless otherwise specified)

  * HIV-1,2 antigen and antibody negative
  * HBsAg negative (chronic hepatitis B carriers without clinical evidence of liver disease can be considered on an individual basis if it is determined that the added risk is justified by the prognosis and lack of treatment alternatives)
  * Hepatitis C antibody negative (positive antibody allowed if antigen (RNA)-negative and no clinical evidence of cirrhosis)
  * Cytomegalovirus (CMV), hepatitis B, Human T-lymphotropic virus (HTLV)-1,2, Epstein-Barr virus (EBV), and Herpes antibody status known
  * Pregnancy test negative (women of childbearing potential only)
* No life-threatening organ dysfunction.

  * Uncontrolled or severe cardiovascular disease, including recent (<6 months) myocardial infarction, angina (symptomatic despite optimal medical management), life-threatening arrhythmia or hypertension
* Able to give informed consent

Exclusion Criteria:

* Women who are of child bearing potential must have a negative pregnancy test (serum pregnancy test - human chorionic gonadotrophin (HCG)) within 48 hours of initiating total body irradiation and agree to use reliable contraception for 1 year following transplant.
* Concomitant severe diseases (respiratory, renal, liver, cardiac failures, psychiatric disorders, neoplasms)
* Recurrent urinary, pulmonary infections.
* Active bacterial, viral, or fungal infection
* Active peptic ulcer disease
* Previous treatments with total lymphoid irradiation or total body irradiation
* Interferon-neutralizing antibody positive with a titer greater than 20
* Relapse in the month preceding enrollment
* Poor compliance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Stem cell engraftment | One month to three years

SECONDARY OUTCOMES:
Disease remission | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.

IPD SHARING:
Plan to Share IPD: Undecided